CLINICAL TRIAL: NCT03389412
Title: The Effect of Clinical Characterization of Children With Monosymptomatic Nocturnal Enuresis on the Efficacy of Desmopressin and Alarm Therapy.
Brief Title: The Effect of Selecting Treatment With Desmopressin or Alarm to Children With Enuresis Based on Home Recordings.
Acronym: DRYCHILD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University Ghent (Other); First Affiliated Hospital of Zhengzhou University, China (Unknown); University Clinical Centre in Gdansk, Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRYCHILD
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Enuresis, Nocturnal
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin; Freezing

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study
Who Masked: Participant
Masking Description: The children and the parents will not know, if there treatment is based on home recordings or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment without evaluating the home recordings, medicin. (Experimental): Children will receive desmopressin without evaluating the home recordings.
  Interventions: Drug: Desmopressin
- Treatment without evaluating the home recordings, alarm. (Experimental): Children will receive conditional alarm without evaluating the home recordings.
  Interventions: Device: Conditional alarm
- Treatment based on home recordings, polyuria. (Active Comparator): Children with polyuria based on the home recordings will receive desmopressin.
  Interventions: Drug: Desmopressin
- Treatment based on home recordings, reduced bladder capacity. (Active Comparator): Children with reduced bladder capacity based on the home recordings will receive the conditional alarm.
  Interventions: Device: Conditional alarm
- Treatment based on home recordings, both. (Active Comparator): Children with polyuria and reduced bladder capacity based on the home recordings will receive desmopressin and the conditional alarm.
  Interventions: Drug: Desmopressin; Device: Conditional alarm
- Treatment based on home recordings, none. (Active Comparator): Children with neither nocturnal polyuria nor reduced bladder capacity based on the home recordings will be randomized to either desmopressin or alarm treatment. If there is no effect of the treatment, the treatment can be switched.
  Interventions: Drug: Desmopressin; Device: Conditional alarm

INTERVENTIONS:
Drug: Desmopressin — The children will be treated with 120 microgram/day the first two weeks. If the child is not completely dry, the dose will be increased to 240 microgram/day the rest of the study period (maximum eight weeks of treatment).
  Other Names: Minirin, melt
  Arms: Treatment based on home recordings, both.; Treatment based on home recordings, none.; Treatment based on home recordings, polyuria.; Treatment without evaluating the home recordings, medicin.
Device: Conditional alarm — Eight weeks of treatment.
  Arms: Treatment based on home recordings, both.; Treatment based on home recordings, none.; Treatment based on home recordings, reduced bladder capacity.; Treatment without evaluating the home recordings, alarm.

SUMMARY:
The aim of this study is to investigate the importance of clinical characterization of children with monosymptomatic nocturnal enuresis (MNE) in order to improve treatment efficacy.

The hypothesis is that clinical characterization by measurement of nocturnal urine production and maximal voided volumes in children with MNE and subsequent treatment tailoring improves the response to first-line treatment approach.

DETAILED DESCRIPTION:
This is a randomized, controlled study.

This study will be performed at Aarhus University Hospital (Denmark), Ghent University Hospital (Belgium) and Hospital of Zhengzhou University (China) following the same protocol.

According to the initial randomization, children will be allocated to treatment without (group A) or with (group B) prior clinical characterization based on home recordings.

Group A: The children will be randomized to either an enuresis alarm or desmopressin without evaluating the home recordings.

Group B: The home recordings will be evaluated and treatment will be based on the recordings. Desmopressin will be administered to the children with nocturnal polyuria and the conditional alarm to the children with reduced bladder capacity. Children with nocturnal polyuria and reduced bladder capacity will be treated with both desmopressin and conditional alarm. Children with neither nocturnal polyuria nor reduced bladder capacity will again be randomized to either desmopressin or alarm treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-14 years.
* Three or more wet nights per week regarding the home registrations.

Exclusion Criteria:

* Ongoing constipation and/or faecal incontinence.
* Daytime symptoms such as urgency, frequency or incontinence.
* Recurrent urinary tract infections.
* Anamnestic, clinical or laboratory findings that can be related to diseases or conditions that might affect the parameters investigated.
* Neurological and/or known clinically significant anatomical abnormalities of the urinary tract.
* Former operations in the urinary tract.
* Prior or ongoing treatment with alarm, desmopressin or anticholinergics.
* Ongoing medication that may interfere with the parameters tested.
* Pregnant or lactating girl.
* Contra-indications for the use of desmopressin: habitual or psychogenic polydipsia, use of diuretics, renal insufficiency, hyponatremia or SIADH.
* Hypersensitivity / allergy to substances in the tablets.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
The number of children who responded to the treatment | Eight weeks
  Evaluated by home recordings
The number of children achieving complete dryness (complete responders) | Eight weeks
  Evaluated by home recordings

SECONDARY OUTCOMES:
Change in wet nights | Eight weeks
  Evaluated by home recordings

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (2):
  - Algemeen Ziekenhuis Sint-Jan Brugge, Bruges
  - Ghent University Hospital, Ghent
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China
- Denmark (2):
  - Aalborg University Hospital, Aalborg, Jylland
  - Aarhus University Hospital, Aarhus, Jylland
- University Clinical Centre in Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hahn D, Stewart F, Raman G. Desmopressin for nocturnal enuresis in children. Cochrane Database Syst Rev. 2025 Jul 29;7(7):CD002112. doi: 10.1002/14651858.CD002112.pub2. PMID 40728007
- [Derived] Jorgensen CS, Dossche L, Zhai R, Maternik M, Kamperis K, Breinbjerg AS, Karamaria S, Thorsteinsson K, Borg B, Wang Y, Li S, Raes A, Wei L, Zurowska A, Hagstrom S, Walle JV, Guo WJ, Rittig S. Development of a Novel Prediction Tool for Response to First-Line Treatments of Monosymptomatic Nocturnal Enuresis: A Randomized, Controlled, International, Multicenter Study (DRYCHILD). J Urol. 2024 Oct;212(4):539-549. doi: 10.1097/JU.0000000000004129. Epub 2024 Jul 1. PMID 38950376